CLINICAL TRIAL: NCT06529328
Title: Effect of Core Stability Exercise Versus Trunk Stabilization Exercise on Balance and Walking Abilities in Cerebral Palsy.
Brief Title: Trunk Stabilization vs. Core Stability Exercises: Impact on Balance and Walking Ability in Cerebral Palsy.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0794
Record Dates: First submitted 2024-06-11; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy,; Balance,; Core Stability,; Trunk Stabilization.
MeSH Terms: conditions — Cerebral Palsy | interventions — Core Stability

STUDY DESIGN:
Intervention Model Description: It will be randomized control trail in which nonprobability convenient sampling will be used. two groups of 2 to 7 years age will be formed in which participants will be randomly divided. Group A: will receive , CP children will receive core stability exercises.
  Group B: Experiment group B, CP children will receive trunk stability exercise.
Who Masked: Participant
Masking Description: participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): For eight weeks, the experimental group in this study will engage in three sessions of thirty to forty-five minutes each, dedicated to core stability exercises that will challenge the muscles of the trunk and abdomen.
  Interventions: Other: core stability
- Group B (Experimental): In addition to receiving 25 minutes of conventional therapy, the subjects participated in a 30-minute trunk stabilization exercise program three days a week on non-consecutive days.
  All tense muscles, including the hamstrings and calf muscles in the lower limb, can benefit from passive stretching exercises. First, it is done five times, then you work your way up to ten repetitions, stretch five times, and finally take five minutes to relax. Extensor muscle strengthening exercises for the back, hips, and knees (for 10 minutes).
  Interventions: Other: core stability

INTERVENTIONS:
Other: core stability — In this study the experimental group will perform core stability exercises 3 times per week for an 8-week period and each session of 30 to 45 minutes, the core stability exercises will work on abdominals and trunk muscles with challenges.Subjects received 25 min conventional therapy in addition to 30 30-minute trunk stabilization exercise program conducted for 3 days\week on non-consecutive days.
  Passive stretching exercises are applied to all tight muscles, including the hamstrings and calf muscles in the lower limb. It is performed five times initially, building up to ten repetitions, stretching for 5 times, and then allowing relaxation for 5time. Strengthening exercises for back, hip, and knee extensor muscles (for 10 minutes).
  Other Names: trunk stability

SUMMARY:
Brain lesions cause cerebral palsy, a chronic condition that affects movement, posture, and balance. Its causes range in age from pregnancy to postpartum, and they can impact the neurological, musculoskeletal, and sensory systems. This causes problems with balance, movement, and posture. It is essential to intervene early for improved life quality. Maintaining a constant center of gravity within your support base is referred to as balance. Walking is putting one foot on the ground at all times and lifting and lowering each foot in turn. The stability of the trunk and core is necessary for muscle coordination and deliberate motions. A study compares the efficiency of trunk stabilization and core exercises to enhance balance and evaluates mobility changes, such as altered muscle strength, endurance, and gait, as a result of two treatment approaches.

DETAILED DESCRIPTION:
Experiment group 1: During the course of the study, the experimental group will engage in three sessions of thirty to forty-five minutes each, dedicated to performing core stability exercises. The exercises will target the challenging muscles of the trunk and abdomen.

Weeks one and two:

* Lying supine and contracting abdominal muscles three sets of twenty repetitions each.
* While lying prone, contract your abdominal muscles three sets of twenty repetitions each.
* Squatting and contracting abdominal muscles for three sets of twenty repetitions each.

Week three: Contracting abdominal muscles while lying supine with one leg extended and the other pressed against the abdomen and bent at the knee Fourth week: ● Pulling the limbs upward while keeping the arms and legs close together and contracting the abdominal muscles (3 sets and 20 reps in each set).

* One leg is raised and pulled outward and backward while performing a squat (3 sets per leg, 20 reps per set).
* Rotate your hips while gripping weights in each hand. Perform three sets of 20 repetitions for each body part.

Fifth week: (3 sets of 10 seconds) holding the abdomen in while sitting on a Swiss ball.

● Squatting with the Swiss ball resting on your shoulder, three sets of fifteen repetitions each.

Elevating both the arms and legs in the prone position at the same time (3 sets and 10 repetitions).

Week six: ● Bending 45 degrees to the left or right. ● Bridging with one leg raised and shoulders and hands on the floor (three sets with a 15-second break in between each set).

● Contracting abdominal muscles on the Swiss ball while lying supine (3 sets, 20 reps per set).

During the seventh week, perform three sets of fifteen reps each of lying supine on a Swiss ball and rotating your trunk to the sides.

* Performing the aforementioned exercise while gripping weights for three sets of fifteen repetitions each.
* Side-lying bridge with leg raises (6 reps on each side of the body, followed by a 10-second rest).

Week eight: ● Lying flat on the Swiss ball with the abdomen tucked in and raising one leg (three sets of twenty repetitions each).

● While squatting, raise the opposing arm and leg three times, completing 20 repetitions per set. - Bridge for three sets, pausing for 15 seconds in between each set, with feet on the Swiss ball and one leg raised.

Experiment group 2: For three days per week on non-consecutive days, the subjects underwent a 30-minute trunk stabilization exercise program in addition to 25 minutes of conventional therapy.

All tense muscles, including the hamstrings and calf muscles in the lower limb, can benefit from passive stretching exercises. First, it is done five times, then you work your way up to ten repetitions, stretch five times, and finally take five minutes to relax. Extensor muscle strengthening exercises for the back, hips, and knees (for 10 minutes).

Next, carry out the exercise for trunk stabilization. The supine exercise involves the child pulling in their abdominals towards their back while lying supine and flexing their knees. Alternatively, the child can place their feet on the dome and lift their legs.

ELIGIBILITY:
Inclusion Criteria:

* ● Gender: both girls and boys;
* ● Age: 2-7 years.
* ● Diagnosis: spastic CP.
* ● According to the modified Ashworth scale, the affected lower extremity's degree of spasticity falls between grades 1 and 2.
* PBS > 32.

Exclusion Criteria:

* ● Got a timing injection with botulinum toxin.
* ● Epilepsy | Seizures.
* ● Lower limb surgery performed throughout the research period.
* Any deformity or orthopedic condition that affects balance. Deficits in vision and hearing with a MACS score higher than three will not be considered.
* ● PBS rating less than 32.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Pediatric Reach Test (Pediatric Functional Reach Test) | 8weeks
  Functional Reach will be measured
Manual Ability Classification System | 8weeks
  ability of children with cerebral palsy to handle objects with the help of their hands.

CONTACTS AND LOCATIONS:
Overall Officials: Saba Munir, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International university, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vitrikas K, Dalton H, Breish D. Cerebral Palsy: An Overview. Am Fam Physician. 2020 Feb 15;101(4):213-220. PMID 32053326